CLINICAL TRIAL: NCT07257120
Title: A Phase IV, Open-label, Single-group Study Evaluating KarXT Concentrations in the Breast Milk and Plasma of Healthy Lactating Female Participants
Brief Title: KarXT Concentrations in the Breast Milk and Plasma of Lactating Females
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0067
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteer; Pharmacokinetics; BMS-986510; KarXT; Cobenfy; Healthy lactating women
MeSH Terms: interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline/trospium chloride

INTERVENTIONS:
Drug: Xanomeline/trospium chloride — Specified dose on specified days
  Other Names: KarXT; BMS-986510

SUMMARY:
The purpose of this study is to characterize the PK of xanomeline and trospium in breast milk and plasma in healthy lactating female participants, following multiple oral administration of KarXT in healthy lactating participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants should have a body mass index (BMI) of 18.0 kg/m2 to 35.0 kg/m2, inclusive, and body weight ≥ 50 kg (110 lb), at screening.
* Participants should have well-established lactation (ie, at least 4 weeks postpartum) and can produce stable milk product (ie, approximately 3 oz per 3 hours at screening) using the methods required for the study.
* Participants should be willing to exclusively pump breast milk throughout the treatment period and during the 24-hour post last dose period of milk collection during the CRU domincile period.
* Participants should agree not to breastfeed or provide milk to infant until after 96 hours post last dose.

Exclusion Criteria:

* Participants must not have evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, 12-lead ECG, or clinical laboratory determinations beyond what is consistent with the target population reference ranges as assessed by the investigator.
* Participants must not have history or presence of clinically significant cardiovascular, pulmonary, renal, hematologic, gastrointestinal (eg, obstructive disorders [including conditions that may decrease GI motility, such as ulcerative colitis, intestinal atony, and myasthenia gravis]), endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the participant or the validity of the study results.
* Other protocol defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of KarXT in Milk | Up to Day 7
Time of maximum observed concentration (Tmax) of KarXT in Milk | Up to Day 7
Area under the concentration-time curve from time zero to 12 hours post morning dose [AUC(0-12)] of KarXT in Milk | Up to Day 7
Area under the concentration-time curve from time zero to 24 hours post morning dose [AUC(0-24)] of KarXT in Milk | Up to Day 7
Average concentration (Cavg) of KarXT in Milk | Up to Day 7
Amount of KarXT recovered in milk within 12 hours of dosing [AR(12)] | Up to Day 7
Total amount of KarXT recovered in milk (AR) | Up to Day 7
Milk-plasma ratio of KarXT (M/P) | Up to Day 7
  Calculated as milk AUC(0-12)/plasma AUC(0-12)

SECONDARY OUTCOMES:
Cmax of KarXT in plasma | Up to Day 7
Tmax of KarXT in plasma | Up to Day 7
AUC (0-12) of KarXT in plasma | Up to Day 7
AUC (0-24) of KarXT in plasma | Up to Day 7
Cavg of KarXT in plasma | Up to Day 7
Estimated daily infant dosage of KarXT | Up to Day 7
Relative infant dosage of KarXT | Up to Day 7
Number of participants with Adverse Events (AEs) | Up to Day 34
Number of participants with Serious Adverse Events (SAEs) | Up to Day 34
Number of participants with physical examination abnormalities | Up to Day 7
Number of participants with vital signs abnormalities | Up to Day 7
Number of participants with 12-Lead electrocardiogram (ECG) abnormalities | Up to Day 7
Number of participants with clinical laboratory abnormalities | Up to Day 7
Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 7
Number of participants with Adverse Events of Special Interest (AESIs) | Up to Day 34

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD | Las Vegas Clinical Research Unit, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07257120.html